CLINICAL TRIAL: NCT02643173
Title: Hepatocellular Carcinoma Recurrence and Anesthesia
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Hyo-Seok Na, Dr, Seoul National University Bundang Hospital
Other Study IDs: HCC recurrence
Record Dates: First submitted 2015-12-29; First posted 2015-12-31 (Estimated); Last update posted 2019-11-22 (Actual); Status verified 2019-11

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Anesthetics, Intravenous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (2):
- Volatile: The investigators retrospectively reviewed and analyzed the electrical medical records of patients who underwent surgery for HCC under the general anesthesia using volatile anesthetics as maintenance agents.
  Interventions: Other: Volatile anesthetics
- Intravenous: The investigators retrospectively reviewed and analyzed the electrical medical records of patients who underwent surgery for HCC under the general anesthesia using intravenous anesthetics as maintenance agents.
  Interventions: Other: Intravenous anesthetics

INTERVENTIONS:
Other: Volatile anesthetics
  Groups: Volatile
Other: Intravenous anesthetics
  Groups: Intravenous

SUMMARY:
The investigators will verify the prognosis of hepatocellular carcinoma (HCC) according to the main anesthetic agents used for the general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing surgery due to the HCC.

Exclusion Criteria:

* Patients undergoing re-operation due to the HCC.
* Patients presenting distant metastasis.
* Patients undergoing liver transplantation surgery.

Ages: 20 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing surgery due to the HCC.
Sampling Method: Non-Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2015-09; Primary Completion 2019-06 (Actual); Study Completion 2019-06 (Actual)

PRIMARY OUTCOMES:
Recurrence of HCC | Postoperative 2 year

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea